CLINICAL TRIAL: NCT03843905
Title: Predictive Value of Innovative Prognostic Markers (Gut Microbiota, Sarcopenia, Metabolic Syndrome and Obesity) on Surgical and Oncologic Results in the Management of Sporadic Colorectal Adenocarcinoma.
Acronym: METABIOTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: M2iSH laboratory (Other); Benoit Chassaing (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-424; 2018-A00352-53 (Other: 2018-A00352-53)
Record Dates: First submitted 2019-02-01; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Neoplasms; Microbiota; Prognosis; Metabolic Syndrome; Sarcopenia
Keywords: Gut microbiota; Colorectal cancer; Sarcopenia; Metabolic syndrome; Prognostic factors; Pathogenic E.coli
MeSH Terms: conditions — Colorectal Neoplasms; Metabolic Syndrome; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — The aim of this translational research project is to study the impact of these new prognostic tools on surgical and oncologic results in a prospective cohort of patients who underwent CRC surgery at the Digestive Surgery Department of the University Hospital of Clermont-Ferrand (France)

SUMMARY:
Colorectal cancer (CRC), second leading cause of cancer worldwide, is associated with a poor prognosis, especially in patients with advanced disease. Therefore, there is still a need to develop new prognostic tools to replace or supplement those routinely used, with the aim to optimize treatment strategies.

Studies on gut microbiota composition provide new strategies to identify powerful biomarkers. Indeed, beyond its beneficial functions for the host, increasing evidences suggest that gut microbiota is a key factor involved in CRC carcinogenesis. Many clinical studies have described an imbalance in the gut microbiota (dysbiosis) in CRC patients, with the emergence of pathogenic bacterial species, Recent studies reported that pks-positive E. coli, a pathogenic bacterial producing toxin encoded by the pks genomic island, is more frequently detected in CRC patients, suggesting a possible role in tumor development. Therefore, this suggests the potential use of microbial signatures associated with CRC for prognostic assessment. Furthermore, influence of body composition profile (BMI, sarcopenia, metabolic syndrome) also appears to be a new relevant prognostic tool regarding surgical and oncological outcomes following CRC surgery.

The aim of this translational research project is to study the impact of these new prognostic tools on surgical and oncologic results in a prospective cohort of patients who underwent CRC surgery at the Digestive Surgery Department of the University Hospital of Clermont-Ferrand (France). This could allow to optimize treatment strategies and provide new ways to identify news promising biomarkers associations in order to better define high risk patients. Investigators aim to identify specific microbial signatures associated with some metabolic profiles in order to improve surgical morbidity and/or response to cancer therapies.

DETAILED DESCRIPTION:
The METABIOTE study will be systematically proposed to patients selected for sporadic CRC surgery during the first preoperative outpatient visit. The attending surgeon will double-check all inclusion and exclusion criteria. An oral and written information will be given to patients, presenting the study.

Then, the following data will be collected propectively:

* Socio-demographic and medical data (personal and familial medical history, current treatments, comorbidities, allergies, Body Mass Index (BMI), ASA score…)
* Blood tests results, including nutritional, hepatic assessment and exploration of a lipidic abnormality.
* Body composition profile: Metabolic syndrome screening, BMI, waist circumference, sarcopenia (skeletal muscle index calculation on CT scan).
* Thoraco-abdomino-pelvic CT scan: sarcopenia, hepatic and splenic density, thanks to a dedicated software (Slice-O-Matic).

Following surgery will be collected :

* Pathological data (TNM stage, MSI, RAS and BRAF status…)
* Surgical results (30-day postoperative medical and surgical morbidity and 90-day postoperative mortality)
* Oncologic results (Overall survival, Disease free survival…)
* Metabolic profile evolution: sarcopenia (SMI), BMI and waist circumference after 3, 6, 12 and 36 months, postoperatively.

Intraoperatively, samples of peritumoral mucosa and tumor specimen and rectal stools will be frozen (-80°) and moved to the research unit for microbiota analysis. Interest bacteria will be grown on selective gelosis and pathogenic E coli will be identified using PCR as well as other specific bacteria involved in CRC. Moreover, global microbiota modifications will be observed using high-throughput sequencing of the bacterial 16S rRNA gene. These data will be associated with body composition profile, clinical data, surgical and oncologic results, and pathological data thanks to a multivariate analysis.

The patients will be monitored according to the Digestive Oncology french recommendations (TNCD).

ELIGIBILITY:
Inclusion Criteria:

* - Male or female, age > to 18 years.
* Histologically proven colonic or high rectal adenocarcinoma
* Absence of metastasis (CT scan) in exams performed preoperatively
* No history of other tumors
* Patients for whom the social and psychological status, the general condition are able to be monitored and/or compliant with the requirements of the study
* Signed and dated informed consent document

Exclusion Criteria:

* - < 18 years, patient in legal incapacity (person deprived of liberty or under guardianship).
* Antibiotic administration within the 2 months before surgery
* Long-term probiotic oral intake
* Inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* Preoperative bowel preparation (oral or rectal) inclued antibiotic and/or antiseptic preparation.
* Metastatic disease
* Genetic CRC : familial adenomatous polyposis, hereditary non polyposis colorectal cancers (HNPCC).
* Patient requiring preoperative radio-chemotherapy or chemotherapy alone
* Medical history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Histologically proven colonic or high rectal adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | at 5 years
  defined by the time between surgery and last follow-up. The 5 years overall survival will be recorded.

SECONDARY OUTCOMES:
Overall survival related to CRC | at 1, 3 and 5 years
  time between surgery and last follow-up. The1-3- and 5 years overall survivals will be recorded
Disease free survival (DFS) | at 1, 3 and 5 years
  time between surgery and first identified recurrence. The1-3- and 5 years disease-free survivals will be recorded
post-operative morbidity | at 30 days
  incidence of postoperative complications (medical and surgical) according to the Clavien-Dindo classification occurring during the hospital stay and up-to 30-day after surgery will be recorded from the audit database
length of hospital stay | at 3 months
  length of hospital stay includes length of stay in Intensive Care unit and Conventional Hospital Unit.
postoperative mortality | at 90 days
  postoperative death until 90 days after surgery
evolution of sarcopenia | at 3,6, 12 and 36 months
  evolution of skeletal muscle index (SMI) identified from pretreatment and oncology follow-up computed tomography scans
evolution Body Mass Index (BMI) | at 3,6,12 and 36 months
  evolution Body Mass Index (BMI) defined during postoperative oncologic follow up clinical consultations (weight measurement)
Microbiota composition | during surgery
  composition of the microbiota according to the sampling site (stools, Peritumoral mucosa and tumor)

CONTACTS AND LOCATIONS:
Overall Officials: Julie VEZIANT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Veziant J, Poirot K, Chevarin C, Cassagnes L, Sauvanet P, Chassaing B, Robin F, Godfraind C, Barnich N, Pezet D, Pereira B, Gagniere J, Bonnet M. Prognostic value of a combination of innovative factors (gut microbiota, sarcopenia, obesity, metabolic syndrome) to predict surgical/oncologic outcomes following surgery for sporadic colorectal cancer: a prospective cohort study protocol (METABIOTE). BMJ Open. 2020 Jan 7;10(1):e031472. doi: 10.1136/bmjopen-2019-031472. PMID 31915159